CLINICAL TRIAL: NCT02144935
Title: Collaborative Assessment of Pediatric Transverse Myelitis: Understand, Reveal, Educate or CAPTURE Study
Acronym: TMCAPTURE
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Benjamin Greenberg, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: 012014-077; 012014-077 (Other: UTSW IRB)
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Myelitis, Transverse; Flaccid Paraplegia, Complete, Acute; Flaccid Paraplegia, Incomplete, Acute
Keywords: pediatrics
MeSH Terms: conditions — Myelitis, Transverse; Paraplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- myelitis, transverse or acute flaccid myelitis: Observational study with online survey participation highlighting outcomes recovery. The surveys can be completed by the child and parent, or if too young to participate, parent only. The survey asks how the child is doing after hospitalization within 6 months of diagnosis, and every 4 months until study end in 2024.

SUMMARY:
Patients and families are invited to participate in an online registry and data repository specifically for patients with transverse myelitis (TM) or acute flaccid myelitis (AFM). The data generated in this study will come from surveys, interviews, review of medical records.

Data from this study will be utilized to guide future clinical trials for children with an acute case of TM or AFM. Parents and school aged children will complete an online survey 7 banks of questions. Each bundle of survey topics have 7-10 questions. We will have both the parent and child complete a outcomes based survey within 6 months of diagnosis and invite to participate every 4 months until study end in 2024.

DETAILED DESCRIPTION:
Both parent and child will participate in the online questionnaires. The validated questionnaires, PROMIS or Patient-Reported Outcomes Measurement Information System, are blocks of 8-10 questions. 7 blocks of questions for the parent and 7 similar blocks for the child: anxiety, depressive symptoms, fatigue, mobility, pain interference, peer relationships, upper extremity function.

Participation via the Internet: When a child or family enters the Transverse Myelitis Association (TMA) website, they will be directed to information about the CAPTURE study. If the family is interested in participation, the TMA will give them the UT southwestern in Dallas, TX research coordinator information. It is up to the parent/guardian to contact the study staff from University Texas Southwestern. Once initial contact is complete, at the family's request, study staff will send the consent form to the interested family. The family will need to email or mail the consent back. Once the signed consent form is in hand, we will send the research survey to the email the parent provides. One survey for the parent, a separate but similar survey for a school aged child.

We will invite parents of school aged children to complete a school survey. This is a one time only questionnaire. Ideally, the parents will complete this either 6 months or 1 year into their child's recovery of TM/AFM.

We invite families living outside of North America to participate in the online survey. They need to be fluent in English, same as the North American cohort.

ELIGIBILITY:
Inclusion Criteria for the registry:

* Diagnosis of transverse myelitis (TM) or acute flaccid myelitis (AFM)
* Patient is within 6 months of symptom onset
* Ability of patent or legal guardian is able to provide informed consent
* Ability of a child 10 or older able to provide assent
* Access to the internet

Exclusion Criteria for the registry:

* Inability to provide appropriate consent or assent
* Diagnosis of multiple sclerosis, neuromyelitis optica, or neuromyelitis optica spectrum disorder

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Transverse Myelitis. Pediatric Acute Flaccid Myelitis. The diagnosis of TM or AFM needs to be within 6 months of symptom onset at the time of consent.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-05; Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Patient and parent reported symptoms of recovery | up to one year post symptom onset
  each parent /guardian and child will fill out a questionnaire examining how you feel about your ability to move and your emotions. This is completed at 3,6,and 12 months after symptoms are diagnosed.

SECONDARY OUTCOMES:
ASIA scale | up to one year after symptom diagnosis
  We will measure the motor (movement) and sensory (touch) of the child above and below the spinal lesion. This is completed at 3 time points 3,6,and 12 months post symptom onset. For the secondary outcomes, the family needs to be able to travel to 1 of the 5 centers listed in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, MD, Principal Investigator — UT Southwestern
Locations (1):
- UTexasSouthwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Transverse Myelitis Association — http://www.myelitis.org